CLINICAL TRIAL: NCT04291911
Title: Prospective Multicentre Observational Study on the Incidence of Hyperoxia in Non-intubated Patients in Intensive Care in Belgium Study OxSIZgen
Brief Title: Retrospective Multicentre Observational Study on the Incidence of Hyperoxia in Non-intubated Patients in Intensive Care in Belgium Study OxSIZgen
Acronym: OxSIZgen
Status: Completed | Type: Observational
Sponsor: SIZ Nursing (Other)
Responsible Party: Principal Investigator, Arnaud Bruyneel, President of SIZ Nursing, RN, CCRN, PhDc, SIZ Nursing
Other Study IDs: SIZNursing
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Hyperoxia
MeSH Terms: conditions — Hyperoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- INTENSIVE CARE UNITS

SUMMARY:
Oxygen is the most widely prescribed therapy in the ICU (intensive care unit) and can save lives in critical patients. While the deleterious effects of hypoxia are apparent and must be actively avoided, hyperoxia also has adverse effects. These include systemic, coronary and cerebral vasoconstriction; decreased coronary blood flow; pulmonary atelectasis and increased free radicals. Despite these deleterious effects, hyperoxia is common and frequent in the ICU (from 22% to 74%).

A recent meta-analysis published in "The Lancet" with more than 16,000 patients demonstrated an association between liberal oxygen therapy and mortality in critical patients. Other meta-analyses confirm its results with high quality data according to the authors.

A randomized controlled trial published in "The New England Journal of Medicine" comparing liberal versus conservative oxygen therapy showed no difference in mechanical ventilation days and mortality (The ICU-ROX, 2019). However, the difference in PaO2 between the two groups was very small and the PaO2 in the liberal group did not exceed 100 mmHg. In any case, conservative oxygen therapy is safe for critical patients.

The recommendations therefore recommend an oxygen saturation between 94-97% in critical patients and 88-92% in patients with COPD (Chronic Obstructive Pulmonary Disease) .

However, to our knowledge, no study has described the incidence of hyperoxia in non-intubated patients in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Patient having oxygen
* Not to be ventilated
* Being over 18 years old

Exclusion Criteria:

* Sickle cell disease patient
* Patient with pneumo/hemothorax
* Pregnant women, prisoners, denial of informed consent
* Patients who are related to an investigator
* Patients undergoing hyperbaric chamber therapy
* Patients with CO
* Patients on ECMO
* Patients with paracoate poisoning...
* Patients included in other interventional studies

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Oxygen patients in intensive care hospitals and no-intubated
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
INCIDENCE HYPEROXIA | one week

CONTACTS AND LOCATIONS:
Locations (1):
- Bruyneel Arnaud, La Louvière, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suzuki S, Mihara Y, Hikasa Y, Okahara S, Ishihara T, Shintani A, Morimatsu H, Sato A, Kusume S, Hidaka H, Yatsuzuka H, Okawa M, Takatori M, Saeki S, Samuta T, Tokioka H, Kurasako T, Maeda M, Takeuchi M, Hirasaki A, Kitaura M, Kajiki H, Kobayashi O, Katayama H, Nakatsuka H, Mizobuchi S, Sugimoto S, Yokoyama M, Kusudo K, Shiraishi K, Iwaki T, Komatsu T, Hirai Y, Sato T, Kimura M, Yasukawa T, Kimura M, Taniguchi M, Shimoda Y, Kobayashi Y, Tsukioki M, Manabe N, Ando E, Kosaka M, Tsukiji T, Tokura C, Asao Y, Sugiyama M, Seto K; Okayama Research Investigation Organizing Network (ORION) investigators. Current Ventilator and Oxygen Management during General Anesthesia: A Multicenter, Cross-sectional Observational Study. Anesthesiology. 2018 Jul;129(1):67-76. doi: 10.1097/ALN.0000000000002181. PMID 29553985
- [Background] Hedenstierna G, Meyhoff CS. Oxygen toxicity in major emergency surgery-anything new? Intensive Care Med. 2019 Dec;45(12):1802-1805. doi: 10.1007/s00134-019-05787-8. Epub 2019 Oct 10. No abstract available. PMID 31599335
- [Background] Asfar P, Singer M, Radermacher P. Understanding the benefits and harms of oxygen therapy. Intensive Care Med. 2015 Jun;41(6):1118-21. doi: 10.1007/s00134-015-3670-z. Epub 2015 Jan 30. No abstract available. PMID 25634474
- [Background] de Graaff AE, Dongelmans DA, Binnekade JM, de Jonge E. Clinicians' response to hyperoxia in ventilated patients in a Dutch ICU depends on the level of FiO2. Intensive Care Med. 2011 Jan;37(1):46-51. doi: 10.1007/s00134-010-2025-z. Epub 2010 Sep 28. PMID 20878146
- [Background] Rachmale S, Li G, Wilson G, Malinchoc M, Gajic O. Practice of excessive F(IO(2)) and effect on pulmonary outcomes in mechanically ventilated patients with acute lung injury. Respir Care. 2012 Nov;57(11):1887-93. doi: 10.4187/respcare.01696. Epub 2012 May 15. PMID 22613692
- [Background] Chu DK, Kim LH, Young PJ, Zamiri N, Almenawer SA, Jaeschke R, Szczeklik W, Schunemann HJ, Neary JD, Alhazzani W. Mortality and morbidity in acutely ill adults treated with liberal versus conservative oxygen therapy (IOTA): a systematic review and meta-analysis. Lancet. 2018 Apr 28;391(10131):1693-1705. doi: 10.1016/S0140-6736(18)30479-3. Epub 2018 Apr 26. PMID 29726345
- [Background] You J, Fan X, Bi X, Xian Y, Xie D, Fan M, Xu W, Zhang K. Association between arterial hyperoxia and mortality in critically ill patients: A systematic review and meta-analysis. J Crit Care. 2018 Oct;47:260-268. doi: 10.1016/j.jcrc.2018.07.014. Epub 2018 Jul 20. PMID 30077082
- [Background] Ni YN, Wang YM, Liang BM, Liang ZA. The effect of hyperoxia on mortality in critically ill patients: a systematic review and meta analysis. BMC Pulm Med. 2019 Feb 26;19(1):53. doi: 10.1186/s12890-019-0810-1. PMID 30808337
- [Background] Stolmeijer R, Bouma HR, Zijlstra JG, Drost-de Klerck AM, Ter Maaten JC, Ligtenberg JJM. A Systematic Review of the Effects of Hyperoxia in Acutely Ill Patients: Should We Aim for Less? Biomed Res Int. 2018 May 14;2018:7841295. doi: 10.1155/2018/7841295. eCollection 2018. PMID 29888278
- [Background] ICU-ROX Investigators and the Australian and New Zealand Intensive Care Society Clinical Trials Group; Mackle D, Bellomo R, Bailey M, Beasley R, Deane A, Eastwood G, Finfer S, Freebairn R, King V, Linke N, Litton E, McArthur C, McGuinness S, Panwar R, Young P; ICU-ROX Investigators the Australian and New Zealand Intensive Care Society Clinical Trials Group. Conservative Oxygen Therapy during Mechanical Ventilation in the ICU. N Engl J Med. 2020 Mar 12;382(11):989-998. doi: 10.1056/NEJMoa1903297. Epub 2019 Oct 14. PMID 31613432
- [Background] O'Driscoll BR, Howard LS, Earis J, Mak V; British Thoracic Society Emergency Oxygen Guideline Group; BTS Emergency Oxygen Guideline Development Group. BTS guideline for oxygen use in adults in healthcare and emergency settings. Thorax. 2017 Jun;72(Suppl 1):ii1-ii90. doi: 10.1136/thoraxjnl-2016-209729. No abstract available. PMID 28507176
- [Background] Siemieniuk RAC, Chu DK, Kim LH, Guell-Rous MR, Alhazzani W, Soccal PM, Karanicolas PJ, Farhoumand PD, Siemieniuk JLK, Satia I, Irusen EM, Refaat MM, Mikita JS, Smith M, Cohen DN, Vandvik PO, Agoritsas T, Lytvyn L, Guyatt GH. Oxygen therapy for acutely ill medical patients: a clinical practice guideline. BMJ. 2018 Oct 24;363:k4169. doi: 10.1136/bmj.k4169. No abstract available. PMID 30355567
- [Background] Perkins GD, Olasveengen TM, Maconochie I, Soar J, Wyllie J, Greif R, Lockey A, Semeraro F, Van de Voorde P, Lott C, Monsieurs KG, Nolan JP; European Resuscitation Council. European Resuscitation Council Guidelines for Resuscitation: 2017 update. Resuscitation. 2018 Feb;123:43-50. doi: 10.1016/j.resuscitation.2017.12.007. Epub 2017 Dec 9. No abstract available. PMID 29233740